CLINICAL TRIAL: NCT02131779
Title: Prostate Cancer Education in African American Churches
Brief Title: Men's Prostate Awareness Church Training
Acronym: M-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 12-0095; American Cancer Society (Other Grant/Funding Number: 119421-RSGT-10-113-01-CPPB)
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer disparities; African American; Spiritually based intervention; Men's Health; Informed Decision Making; Community Based Participatory Research; Health Communication; Health Information Technology; Community Health Advisors
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Co-Educational Workshops (Experimental): Community health advisors will be trained using traditional/classroom methods and provided with technical assistance/support to implement the 4 part health series with men and women dyads. Technical assistance and support will be given as needed to community health advisors. Workshop sessions will include didactic lecture, group discussions, video and group exercises.
  Interventions: Behavioral: Co-Educational Workshops
- Men's Workshops (Active Comparator): Community health advisors will be trained using traditional/classroom methods and provided with technical assistance/support as needed to deliver 4 part educational sessions to men only groups to relay information about making an informed decision about prostate cancer screening. Workshop sessions will include didactic lecture, group discussions, video and group exercises.
  Interventions: Behavioral: Men's Workshops

INTERVENTIONS:
Behavioral: Men's Workshops — Two male Community Health Advisors will be trained using traditional/classroom methods and provided with technical assistance/support to implement the 4 part workshop series.
  Arms: Men's Workshops
Behavioral: Co-Educational Workshops — One male and one female Community Health Advisor will be trained using traditional/classroom methods and provided with technical assistance/support to implement the 4 part workshop series. Two break out sessions will occur in the Health Partner condition with separate discussion sessions for men and female health partners.
  Arms: Co-Educational Workshops

SUMMARY:
The objective of the Prostate Cancer Education in African American Churches project is to develop and evaluate a spiritually-based educational intervention for Informed Decision Making (IDM) for prostate cancer screening to be delivered to African American men in church settings.

DETAILED DESCRIPTION:
The specific aims of the project are to 1) develop, and 2) test the efficacy of a spiritually-based cancer communication intervention to increase IDM for prostate cancer screening among African American men in church settings, and including women as supportive "health partners".

A randomized controlled trial is utilized, in which churches will be randomized to: 1) male-only educational groups; and 2) co-educational groups where women supportive "health partners" are invited to attend with the men in dyads, and then break out into men's and women's discussion groups. These two approaches are compared through use of cluster randomized design to determine whether the addition of the women health partner increases the intervention efficacy in the study outcome of informed decision making for prostate cancer screening.

ELIGIBILITY:
Inclusion Criteria:

Male Study Participants

* African American Men church attending men
* 40-69 years of age Advisory Panel

  * Knowledgeable about the community where the intervention is implemented, adults ages 21+, review materials and provide input for intervention development and program implementation Pastors
  * Willing to conduct the intervention at church
  * Support the program
  * Designate two individuals to serve as community health advisors
  * Identify a ministry in the church which will champion the project Community Health Advisors
  * attend a 6 hour training and 1 hour certification
  * assist in recruitment of study participants
  * recruit up to 24 men
  * recruit up to 24 females to attend sessions with men in 10 Health Partner Churches
  * prepare and conduct the 4 part workshop series
  * serve as liaisons between the project and study team Workshop Participants
  * self-identified, African American men (40-69), Health Partners --over 18 years of age, able to complete self-administered paper-and-pencil surveys

Exclusion Criteria:

* Workshop participants with a history of prostate cancer, do not meet the age criteria

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2012-02; Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Informed Decision making for Prostate Cancer Screening | Baseline to 12 month follow-up
  IDM for prostate cancer screening for African American men participating in a church-based group educational workshops will be measured at baseline and 12 months. Survey assessments items for informed decision making include: stage of decision making, preference for decision making, and self-efficacy for decision making.

SECONDARY OUTCOMES:
Theory-based measures, prostate cancer knowledge, and prostate cancer screening | Change from baseline to 12 month follow-up
  Health Belief Model-based scales including perceived benefits of screening; perceived barriers to screening; self-efficacy for screening; and knowledge including prostate cancer knowledge; knowledge about the prostate cancer screening controversy; and prostate cancer screening through self-report receipt of prostate specific antigen test and digital rectal examination

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Holt, PhD, Principal Investigator — University of Maryland School of Public Health
Locations (1):
- University of Maryland School of Public Health, College Park, Maryland, United States

REFERENCES:
- [Background] Saunders DR, Holt CL, Whitehead TL, Atkinson NL, Le D, Wang MQ, Slade JL, Muwwakkil B, Williams R, Schulz E, Naslund M. Development of the men's prostate awareness church training: church-based workshops for African American men. Fam Community Health. 2013 Jul-Sep;36(3):224-35. doi: 10.1097/FCH.0b013e318292eb40. PMID 23718958
- [Derived] Le D, Holt CL, Saunders DR, Wang MQ, Coriolan A, Savoy AD, Slade JL, Muwwakkil B, Atkinson NL. Feasibility and acceptability of SMS text messaging in a prostate cancer educational intervention for African American men. Health Informatics J. 2016 Dec;22(4):932-947. doi: 10.1177/1460458215598636. Epub 2015 Aug 30. PMID 26324051
- [Derived] Saunders DR, Holt CL, Le D, Slade JL, Muwwakkil B, Savoy A, Williams R, Whitehead TL, Wang MQ, Naslund MJ. Recruitment and Participation of African American Men in Church-Based Health Promotion Workshops. J Community Health. 2015 Dec;40(6):1300-10. doi: 10.1007/s10900-015-0054-9. PMID 26089253
- [Derived] Holt CL, Le D, Saunders DR, Wang MQ, Slade JL, Muwwakkil B, Williams R, Atkinson NL, Whitehead TL, Naslund M. Informed Decision-Making and Satisfaction with a Church-Based Men's Health Workshop Series for African-American Men: Men-Only vs. Mixed-Gender Format. J Cancer Educ. 2015 Sep;30(3):530-4. doi: 10.1007/s13187-014-0731-x. PMID 25330866
- See also: Community Health Awareness, Messages & Prevention --University of Maryland, Research lab where the project is based — https://sph.umd.edu/research-impact/laboratories-projects-and-programs/community-health-awareness-messages-and-prevention-champ-lab
- See also: American Cancer Society — http://www.cancer.org